CLINICAL TRIAL: NCT05998109
Title: PheCheck Feasibility Study
Status: Completed | Type: Observational
Sponsor: Lumos Diagnostics (Industry)
Collaborators: Aptatek Biosciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: CLP-0012
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Phenylketonurias
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: PheCheck™ — Quantitative, single-use, rapid test Intended for home-based self-testing and monitoring of PKU.
  1 fingerstick specimen collected at each study visit
Diagnostic Test: HPLC Amino Acid Analyzer — 1 venous specimen collected at each study visit
Diagnostic Test: Dried Blood Spot Cards — capillary blood specimen collected at each study visit

SUMMARY:
The goal of this feasibility study clinical trial is to compare the accuracy of PheCheck™ for the rapid quantitative detection of phenylalanine (Phe) with the gold standard (HPLC amino acid analyzer), in patients with PKU.

The main aims are:

* Evaluate the accuracy of PheCheck as compared to the gold standard
* Evaluate ease of use by lay participants

DETAILED DESCRIPTION:
The primary objective of this feasibility study is to evaluate the accuracy of the analyte concentration of PheCheck™ for the rapid, quantitative detection of phenylalanine (Phe) from capillary blood compared to the gold standard (HPLC amino acid analyzer) which quantitatively measures Phe in venous blood.

The study will enroll subjects into one study cohort. It will include patients 10 years or older, monitored for Phenylketonuria (PKU), hyperphenylalaninemia or PKU during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* 10 years of age or older
* Being monitored for Phenylketonuria (PKU), hyperphenylalaninemia or for PKU during pregnancy Signed informed consent

Exclusion Criteria:

* Younger than 10 years of age
* Not being monitored for Phenylketonuria (PKU), hyperphenylalaninemia or for PKU during pregnancy
* Lack of signed informed consent
* Previous enrollment in the study and has completed study visit 1 and 2

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients ≥ 10 years who are undergoing monitoring for Phenylketonuria (PKU)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Concentration of phenylalanine (Phe) from PheCheck as compared to HPLC amino acid analyzer | 6-8 weeks
  The primary outcome is the concentration of phenylalanine (Phe) from capillary blood as compared to the gold standard HPLC amino acid analyzer

CONTACTS AND LOCATIONS:
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided